CLINICAL TRIAL: NCT01177852
Title: Multicenter Clinical Trial, Phase III, Controlled, Open, Parallel Group, Randomized, Comparing the Fixed Dose Combination of Diphenhydramine + Dropropizine + Pseudoephedrine and the Combined Use of Dropropizine and Fixed Dose Combination of Pseudoephedrine Hydrochloride + Brompheniramine Maleate Used Orally for Evaluation of Efficacy and Safety in Control Cough and the Relief of Nasal Symptoms in Children 2 to 12 Years Old, Suffering From Non-productive Cough and Acute Rhinitis.
Brief Title: Evaluation of Efficacy and Safety in Control Cough and the Relief of Nasal Symptoms in Children 2-12 Years Old,Suffering From Cough and Acute Rhinitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Carla Rosana Goulart Silva Peron, MD, Ache Laboratorios Farmaceuticos S.A
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-NTS-03(02/10)
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Inflammation; Cough; Rhinitis
Keywords: cough, acute rhinitis, common cold, nasal symptoms, children.; Acute inflammation upper airway
MeSH Terms: conditions — Inflammation; Cough; Rhinitis; Common Cold | interventions — Diphenhydramine; dipropizine; Pseudoephedrine; Brompheniramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Notuss® syrup (Experimental): Group 1: fixed dose combination of diphenhydramine + dropropizine + pseudoephedrine (Notuss® syrup).
  Interventions: Drug: diphenhydramine + dropropizine + pseudoephedrine
- Dropropizine + Pseudoephedrine and brompheniramine (Active Comparator): Group 2: combined use of dropropizine and fixed dose combination of pseudoephedrine hydrochloride + brompheniramine maleate.
  Interventions: Drug: Dropropizine and fixed dose combination of pseudoephedrine hydrochloride + brompheniramine maleate (Dimetapp® elixir).

INTERVENTIONS:
Drug: diphenhydramine + dropropizine + pseudoephedrine — Group 1: fixed dose combination of diphenhydramine + dropropizine + pseudoephedrine (Notuss® syrup).
  Posology: The medicine treat will be as follows:
  - Notuss® syrup Age: 2-5 years / Dosage: 5,0 mL Age: 6-12 years / Dosage: 10,0 ml
  Arms: Notuss® syrup
Drug: Dropropizine and fixed dose combination of pseudoephedrine hydrochloride + brompheniramine maleate (Dimetapp® elixir). — Dropropizine:
  Age: 2 - 3 years / Dosage: 5,0 ml Age: 4 - 12 years / Dosage: 10,0 ml
  Pseudoephedrine hydrochloride + brompheniramine maleate:
  Age: 2 - 3 years / Dosage: 2,5 ml Age: 4 - 6 years / Dosage: 5,0 ml Age: 7 - 9 years / Dosage: 7,5 ml Age: 10 - 12 years / Dosage: 10,0 ml
  Arms: Dropropizine + Pseudoephedrine and brompheniramine

SUMMARY:
Multicenter clinical trial, phase III, controlled by active medicine, open, randomized, enroll 962 children, 2 to 12 years old, that suffer acute inflammation upper airway characterized by non-productive cough, daytime/nighttime, with duration for at least 3 and no more than 5 consecutive days (without systemic/topic use of medication during this period) followed by nasal congestion, with or without associate other nasal symptoms (sneezing, runny nose, nasal itching and/or mouth breathing). The subjects will be allocated in 2 parallel groups, and will receive the medicines of study, according of the randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 2 and 12 years old, of both sexes;
2. Clinical condition compatible with acute rhinitis accompanied by nasal obstruction;
3. Non-productive cough, daytime and/or nighttime with at least 3 and up 5 consecutive days in duration;
4. Score greater than or equal to 3 points on the cough severity score (As per item 4.1.2);
5. Score greater than or equal to 2 points on the nasal obstruction severity score (As per item 4.1.3);
6. ICF signed by a parent/caregiver/representant;
7. Parent/Caregiver/Representant capacity, according to investigator evaluation, for compliance at the treatment and protocol requirements, fulfilling the regular visits;

Exclusion Criteria:

1. Non-productive cough with purulent smear, fever (axillar temperature superior than 37,8°C/100°F), purulent runny nose and other signs and symptoms of bacteria infection of upper and lower airways at 7 days before the screening/randomization visit;
2. Septal deviation level III (in any region and any nasal cavity) and/or nasal polyps or other determinants conditions of nasal congestion;
3. Previous diagnosis of asthma;
4. Patients under treatment for chronic allergy;
5. Presence of purulent or mucopurulent secretion, nasal vault or mal formations (cleft lip or cleft nasolabial corrected or not) in nasal vestibule;
6. Current use of systemic antibiotics for any reason;
7. Use of prohibited medicine within the prescribed period before V0 as shown in item 9.3 of this protocol;
8. Participation in last one year of clinical protocols;
9. Any psychiatric diseases, including major depression;
10. Presence of mental retardation from any cause;
11. Diagnosis of renal or hepatic failure;
12. History of hypersensitivity to any component of the study drugs;
13. Relatives of sponsor´s or study site´s employee;
14. Current evidence of clinically significant diseases: hematopoietic, gastrointestinal, cardiovascular, hepatic, renal, neurological, endocrine, psychiatric, autoimmune, pulmonary, or another disease that block the patient participation;
15. Patient or parent/caregiver/representant with a history of lack of compliance to treatment or previous treatment protocols;
16. Any finding of clinical observation (anamnesis and physical exam) laboratory abnormality (eg, blood glucose, blood count), disease (for example, liver, cardiovascular system, lung) or therapy that, in opinion of the investigator, may endanger the patient or interfere with the endpoints of study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of nasal congestion and cough | Evaluated on the day 2 after beginning treatment
  Participants were evaluated (by a parent/guardian/caregivers) for pain intensity by using a 4-point rating scale: 0=none, 1=mild, 2=moderate, and 3=severe.

SECONDARY OUTCOMES:
Improvement of nasal congestion and cough | Evaluated on the 7(±1) day after beginning treatment
  Participants were evaluated (by a parent/guardian/caregivers) for pain intensity by using a 4-point rating scale: 0=none, 1=mild, 2=moderate, and 3=severe.
Improvement of non-obstructive nasal symptoms | Evaluated on the day 2 and 7 (±1) after beginning treatment
  Participants were evaluated (by a parent/guardian/caregivers for pain intensity by using a sum of 4-point rating scale: 0=none, 1=mild, 2=moderate, and 3=severe.
Reduction of the frequency of nighttime awakenings of parent/guardian/roommate of the child | Evaluated on the day 2 and 7 (±1) after beginning treatment
Reduction of vomiting frequency episodes triggered by coughing | Evaluated on the day 2 and 7 (±1) after beginning treatment
Improvement of acute rhinitis signs | Evaluated on the day 2 and 7 (±1) after beginning treatment
  Assessed by anterior rhinoscopy and application of specific clinical scores
Use of rescue medication | Evaluated on the day 2 and 7 (±1) after beginning treatment
Overall impression of improvement by the investigator | Evaluated on the day 2 and 7 (±1) after beginning treatment
  Specific scale and overall impression of improvement by a parent/guardian/ caregiver of the child
Safety descriptive about occurence of adverse events, evaluation of results of general physical examination. | Will be evaluated during the 7(± 1) days of treatment
  Collection of safety data throughout the whole study period